CLINICAL TRIAL: NCT01687244
Title: A Phase 2, Randomized, Open Label, Parallel Arm Study to Evaluate the Safety and Efficacy of rAd-IFN/Syn3 Following Intravesical Administration in Subjects With High Grade, BCG Refractory or Relapsed Superficial Bladder Cancer
Brief Title: Intravesical Administration of rAd-IFN/Syn3 in Patients With BCG-Refractory or Relapsed Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FKD Therapies Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rAd-IFN-CS-002
Record Dates: First submitted 2012-09-06; First posted 2012-09-18 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Superficial Bladder Cancer
Keywords: BCG Refractory or Relapsed Superficial Bladder Cancer; rAd-IFN; Syn3; Intravesical; transitional cell carcinoma of the bladder; superficial non-muscle invasive tumor; Interferon alpha2b; INSTILADRIN
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant did not know if they received a high or low dose.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rAd-IFN Dose 1x10^11vps/ml (Experimental): Subjects will be randomly assigned to one of two INSTILADRIN arms.
  Interventions: Drug: INSTILADRIN
- rAd-IFN dose 3x10^11 vps/ml (Experimental): Subjects will be randomly assigned to one of two INSTILADRIN arms.
  Interventions: Drug: INSTILADRIN

INTERVENTIONS:
Drug: INSTILADRIN — The INSTILADRIN components will be mixed with a diluent. The total dose will be given as a single, one-hour intravesical administration which may, depending on clinical response, be repeated every 3 months up to a maximum of 4 instillations.
  Other Names: rAd-IFN/Syn3

SUMMARY:
This Phase 2 study is designed to assess the efficacy and safety of INSTILADRIN (rAd-IFN with Syn3) when given intravesically to patients with high grade non-muscle invasive bladder cancer who are refractory to or have relapsed from BCG therapy. The pharmacodynamics of INSTILADRIN will also be studied by measuring the interferon (IFNα2b) levels excreted in the urine. rAd-IFN is a non-replicating recombinant adenovirus type 5 (Ad5)-vector encoding the interferon alpha-2b (IFNα2b) gene. Syn 3 is clinical surfactant excipient which enhances the ability of the adenoviral vector to transfect cells in the bladder wall.

DETAILED DESCRIPTION:
Criteria for Evaluation:

Efficacy: A Response is defined as no evidence of recurrence of a high grade tumor by cystoscopy, cytology or if clinically indicated, biopsy.

Safety: The safety and tolerability of INSTILADRIN will be evaluated based on adverse event reports, vital signs, ECGs, clinical laboratory values and results of physical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older at the time of consent
2. Able to give informed consent
3. Subjects with high grade BCG-refractory or relapsed NMIBC including

   * High grade non-invasive papillary carcinomas (Ta) and subjects with high grade tumors that invade sub-epithelial connective tissue (T1) or
   * Carcinoma in situ (CIS) only or
   * CIS and Ta or T1 tumors Refractory is defined as failure to achieve a disease-free state at six months after adequate induction of BCG therapy with either maintenance or re-induction at 3 months. Adequate induction is defined as a minimum of 5 out of 6 induction doses and adequate maintenance is defined as a minimum of 2 out of 3 doses of treatment.

   Relapse is defined as recurrence within 1 year after a complete response to BCG treatment
4. Complete resection of visible papillary lesions or CIS by TURBT or endoscopic resection between 14 and 60 days prior to beginning study treatment
5. Available for the whole duration of the study
6. Life expectancy >2 years, in the opinion of the investigator
7. ECOG status 2 or less
8. Absence of upper tract urothelial carcinoma
9. Female subjects of childbearing potential must use maximally effective birth control during the period of therapy, must be willing to use contraception for 1 month following the last study drug infusion and must have a negative urine or serum pregnancy test upon entry into this study. Otherwise, female subjects must be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile.
10. Male subjects must be surgically sterile or willing to use a double barrier contraception method upon enrollment, during the course of the study, and for 1 month following the last study drug infusion.
11. Adequate laboratory values.

    * Hemoglobin ≥10 g/dL.
    * WBC ≥4000/μL.
    * ANC ≥2000/μL.
    * Platelet count ≥100,000/μL.
    * INR within institutional normal limits.
    * aPTT within institutional normal limits.
    * AST ≤1.5 x ULN.
    * ALT ≤1.5 x ULN.
    * Total bilirubin within institutional normal limits.
    * Creatinine ≤1.5 x ULN.

Exclusion Criteria:

1. Current or previous evidence of muscle invasive or metastatic disease
2. Current systemic therapy for bladder cancer
3. Current or prior pelvic external beam radiotherapy
4. Prior treatment with adenovirus-based drugs
5. Suspected hypersensitivity to interferon alpha
6. Existing urinary tract infection or bacterial cystitis
7. Clinically significant and unexplained elevated liver or renal function tests
8. Women who are pregnant or lactating
9. Severe cardiovascular disease
10. History of malignancy of other organ system within past 5 years (except treated basal cell carcinoma or squamous cell carcinoma of the skin)
11. Subjects who cannot hold instillation for 1 hour
12. Subjects who cannot tolerate intravesical dosing or intravesical surgical manipulation
13. Intravesical therapy within 6 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dinney, MD, Study Chair — M.D. Anderson Cancer Center

IPD SHARING:
Plan to Share IPD: No
A manuscript will be published on the results of the study

REFERENCES:
- [Derived] Konety BR, Lotan Y, Myers A. Safety of nadofaragene firadenovec-vncg: review of data from phase 2 and phase 3 studies. Can J Urol. 2025 Mar 18;32(1):29-36. doi: 10.32604/cju.2025.064710. PMID 40194933
- [Derived] Shore ND, Boorjian SA, Canter DJ, Ogan K, Karsh LI, Downs TM, Gomella LG, Kamat AM, Lotan Y, Svatek RS, Bivalacqua TJ, Grubb RL 3rd, Krupski TL, Lerner SP, Woods ME, Inman BA, Milowsky MI, Boyd A, Treasure FP, Gregory G, Sawutz DG, Yla-Herttuala S, Parker NR, Dinney CPN. Intravesical rAd-IFNalpha/Syn3 for Patients With High-Grade, Bacillus Calmette-Guerin-Refractory or Relapsed Non-Muscle-Invasive Bladder Cancer: A Phase II Randomized Study. J Clin Oncol. 2017 Oct 20;35(30):3410-3416. doi: 10.1200/JCO.2017.72.3064. Epub 2017 Aug 23. PMID 28834453

RESULTS

PARTICIPANT FLOW:
Groups:
- rAd-IFN Dose 1x10^11vps/ml: Patients were randomized to the 1x10^11vps/ml rAd-IFN/Syn3 arm.
  A 75 mL dose of rAd-IFN/Syn3 was given as a single, one-hour intravesical administration and, depending on clinical response, was repeated every 90 Days up to a maximum of 4 instilations.
- rAd-IFN Dose 3x10^11 Vps/ml: Patients were randomized to the 3x10^11vps/ml rAd-IFN/Syn3 arm.
  A 75 mL dose of rAd-IFN/Syn3 was given as a single, one-hour intravesical administration and, depending on clinical response, was repeated every 90 Days up to a maximum of 4 instilations.
Period: Overall Study
Arm/Group | rAd-IFN Dose 1x10^11vps/ml | rAd-IFN Dose 3x10^11 Vps/ml
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- rAd-IFN Dose 1x10^11vps/ml: Patients were randomly assigned to the 1x10^11vps/ml of rAd-IFN/Syn3 arm.
- rAd-IFN Dose 3x10^11 Vps/ml: Patients were randomly assigned to the 3x10^11vps/ml of rAd-IFN/Syn3 arm.
- Total: Total of all reporting groups
Arm/Group | rAd-IFN Dose 1x10^11vps/ml | rAd-IFN Dose 3x10^11 Vps/ml | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 7 | 9
  >=65 years | 19 | 12 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (8.07) | 71.1 (9.42) | 71.1 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 19 | 14 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Incidence of High Grade-Recurrence Free Survival at 360 Days
Description: Following the initial treatment, patients were clinically evaluated and re-treated at the Days 90, 180, and 270 time points, as outlined below. The decision to repeat treatment was determined by the clinical response observed following the previous treatment(s). Patients were assessed for High-Grade disease recurrence by cytology, cystoscopy and, if clinically indicated, biopsies were performed to obtain accurate staging. If no evidence of recurrence of High-Grade disease was detected, then a further dose of rAd-IFN/Syn3 was administered as maintenance therapy. Patients who had recurrence of High-Grade disease were withdrawn from treatment but were followed for survival and time to cystectomy. At 360 Days, a final efficacy evaluation was performed for patients receiving 4 doses of drug. This included cystoscopy, cytology, and biopsy.
Time Frame: 360 Days
Measure: Count of Participants; unit: Participants
Groups:
- rAd-IFN Dose 1x10^11 Vps/ml: Subjects were randomly assigned to the 1x10^11 vps/mI rAd-IFN/Syn3 arm.
- rAd-IFN Dose 3x10^11vps/ml: Patients were randomly assigned to the 3x10^11vps/ml rAd-IFN/Syn3 arm.
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants | 7 | 7
Statistical Analysis 1: Comparison: rAd-IFN Dose 3x10^11vps/ml; The primary efficacy endpoint was the incidence of high-grade recurrence-free survival at 12 months. The proportion of patients achieving high-grade recurrence-free survival at 12 months was reported for each dose group, together with an exact 90% confidence interval for the proportion; Test type: Superiority or Other; Not applicable: the primary analysis was a calculation of a confidence interval; HGRF survival at 12 months = 33.3, 90% CI 2-sided [16.8 to 53.6]
Statistical Analysis 2: Comparison: rAd-IFN Dose 1x10^11 Vps/ml; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; HGRF survival at 12 months = 36.8, 90% CI 2-sided [18.8 to 58.2] — The proportion of subjects achieving high-grade recurrence-free survival at 12 months

2. Secondary Outcome: Safety of rAd-IFN/Syn3
Description: Treatment Emergent Adverse Events (AEs) for patients receiving study drug were described by NCI-CTCAE V4.03 terminology according to System Organ Class.
Time Frame: 360 Days
Measure: Count of Participants; unit: Participants
Groups:
- rAd-IFN Dose 1x10^11vps/ml: Patients were randomly assigned to the 1x10^11vps/ml rAd-IFN/Syn3 arm.
- rAd-IFN Dose 3x10^11 Vps/ml: Patients were randomly assigned to the 3x10^11 vps/ml rAd-IFN/Syn3 arm.
Arm/Group | rAd-IFN Dose 1x10^11vps/ml | rAd-IFN Dose 3x10^11 Vps/ml
Number analyzed (Participants) | 21 | 19
Participants | 20 | 19

3. Secondary Outcome: Incidence of High Grade Recurrence-Free Survival at 3 Months (90 Days).
Description: All patients were evaluated 3 Months (90 Days) after the start of treatment for recurrence of high grade disease by cytology, cystoscopy, and biopsy if clinically indicated. Patients that we free of High-Grade disease recurrence received another dose. Data are presented as the number and percent of patients with High-Grade disease recurrence.
Time Frame: 90 Days
Population: All patients at 90 Days were assessed for High-Grade disease by cytology, cystoscopy, and biopsy if clinically indicated.
Measure: Count of Participants; unit: Participants
Groups:
- rAd-IFN Dose 1x10^11 Vps/ml: Patients were randomly assigned to the 1x10^11 vps/ml rAd-IFN/Syn3 arm.
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants | 10 | 13

4. Secondary Outcome: Incidence of High Grade-Recurrence-Free Survival at 6 Months (180 Days).
Description: All patients were evaluated 6 Months (180 Days) after the start of treatment for recurrence of high grade disease by cytology, cystoscopy, and biopsy if clinically indicated. Patients that we free of High-Grade disease recurrence received another dose. Data are presented as the number and percent of patients with High-Grade disease recurrence.
Time Frame: 180 Days
Population: All patients receiving a dose at 90 Days were assessed at 180 Days for High-Grade disease by cytology, cystoscopy, and biopsy if clinically indicated.
Measure: Count of Participants; unit: Participants
Groups:
- rAd-IFN Dose 1x10^11 Vps/ml: Patients were randomly assigned to the 1x10^11 vps/ml rAd-IFN/Syn3 arm.
  .
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants | 8 | 9

5. Secondary Outcome: Incidence of High Grade-Recurrence-Free Survival at 9 Months (270 Days).
Description: All patients were evaluated 9 Months (270 Days) after the start of treatment for recurrence of high grade disease by cytology, cystoscopy, and biopsy if clinically indicated. Patients that we free of High-Grade disease recurrence received a final dose. Data are presented as the number and percent of patients with High-Grade disease recurrence.
Time Frame: 270 Days
Population: All patients that received a dose at Day 180 were assessed for High-Grade disease by cytology, cystoscopy, and biopsy if clinically indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants | 8 | 9

6. Secondary Outcome: Incidence of Cystectomy in All Patients
Description: This secondary objective measures the incidence of cystectomy at 360 Days for the Efficacy Analysis Set.
Time Frame: 360 Days
Population: The data are presented as the number of patients per dose group having a cystectomy during the 360 days of the study.
Measure: Count of Participants; unit: Participants
Groups:
- rAd-IFN Dose 1x10^11vps/ml: Patients were randomly assigned to the 1x10^11 vps/ml rAd-IFN/Syn3 arm.
Arm/Group | rAd-IFN Dose 1x10^11vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants | 0 | 0

7. Secondary Outcome: Overall Survival in All Patients.
Description: Overall survival was defined as the number who survived from the first dose of rAd-IFN/Syn3 to the end of the primary assessment (360 Days) or Withdrawal.
Time Frame: 360 Days
Population: The data are presented as the number of patients who survived the study (360 Days). All patients were monitored for this endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- rAd-IFN Dose 1x10^11 Vps/ml: Patients were randomly assigned to the 1x10^11 vps/mI rAd-IFN/Syn3 arm.
- rAd-IFN Dose 3x10^11vps/ml: Subjects were randomly assigned to the 3x10^11vps/ml rAd-IFN/Syn3 arm.
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants | 21 | 19

8. Secondary Outcome: Number of Patients With Elevated Levels of Viral Vector in Blood
Description: The level of viral vector as measured by qPCR in blood was determined in all patients on the initial day of dosing Day 1 (pre-dose) and at Day 2, Day 4, Day 12, and for patients that were free of High-Grade disease recurrence and received a second dose at Day 91 (pre-dose), Day 92, Day 94, and Day 103.
Time Frame: 103 Days
Population: Data are reported as number of patients demonstrating viral vector by qPCR in blood.
Measure: Count of Participants; unit: Participants
Arm/Group | rAd-IFN Dose 1x10^11vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants
  Pre-Dose Day 1 | 0 | 0
  Day 2 | 0 | 0
  Day 4 | 0 | 0
  Day 12 | 0 | 0
  Pre-Dose Day 91: number analyzed (Participants) | 10 | 13
  Pre-Dose Day 91 | 0 | 0
  Day 92: number analyzed (Participants) | 10 | 13
  Day 92 | 0 | 0
  Day 94: number analyzed (Participants) | 10 | 13
  Day 94 | 0 | 0
  Day 103: number analyzed (Participants) | 9 | 12
  Day 103 | 0 | 0

9. Secondary Outcome: Number of Patients With Elevated Levels of Viral Vector in Urine
Description: The level of viral vector as measured by qPCR in urine was determined in all patients on the initial day of dosing Day 1 (pre-dose) and at Day 2, Day 4, Day 12, and for patients that were free of High-Grade disease recurrence and received a second dose at Day 91 (pre-dose), Day 92, Day 94, and Day 103.
Time Frame: 103 Days
Population: Data are reported as number of patients demonstrating increased levels of viral vector by qPCR in urine.
Measure: Count of Participants; unit: Participants
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants
  Pre-Dose Day 1 | 1 | 0
  Day 2: number analyzed (Participants) | 21 | 18
  Day 2 | 21 | 18
  Day 4 | 20 | 19
  Day 12: number analyzed (Participants) | 20 | 19
  Day 12 | 17 | 16
  Pre-Dose Day 91: number analyzed (Participants) | 10 | 13
  Pre-Dose Day 91 | 1 | 2
  Day 92: number analyzed (Participants) | 10 | 11
  Day 92 | 10 | 11
  Day 94: number analyzed (Participants) | 9 | 12
  Day 94 | 8 | 11
  Day 103: number analyzed (Participants) | 8 | 13
  Day 103 | 2 | 4

10. Secondary Outcome: Number of Patients With Elevated IFN alpha2b Protein Levels in Serum
Description: The levels of serum IFN alpha2b protein as measured by ELISA were determined in all patients on the initial day of dosing (Pre-Dose Day 1), at Day 2, Day 4, Day 12, and for patients that were free of High-Grade disease recurrence and received subsequent doses at Day 91 (pre-dose), Day 92, Day 94, Day 103, Day 180 (pre-dose), Day 270 (pre-dose), and Day 360 or Withdrawal.
Time Frame: 360 Days
Population: Data are reported as the number of patients with increased levels of IFN alpha2b protein in serum.
Measure: Count of Participants; unit: Participants
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants
  Pre-Dose Day 1 | 1 | 1
  Day 2: number analyzed (Participants) | 21 | 18
  Day 2 | 2 | 10
  Day 4 | 1 | 6
  Day 12: number analyzed (Participants) | 20 | 19
  Day 12 | 1 | 1
  Day 91: number analyzed (Participants) | 10 | 13
  Day 91 | 1 | 1
  Day 92: number analyzed (Participants) | 10 | 12
  Day 92 | 1 | 1
  Day 94: number analyzed (Participants) | 10 | 11
  Day 94 | 1 | 1
  Day 103: number analyzed (Participants) | 9 | 13
  Day 103 | 1 | 1
  Pre-Dose Day 180: number analyzed (Participants) | 7 | 9
  Pre-Dose Day 180 | 0 | 0
  Pre-Dose Day 270: number analyzed (Participants) | 7 | 9
  Pre-Dose Day 270 | 0 | 0
  Day 360 or Withdrawal: number analyzed (Participants) | 14 | 13
  Day 360 or Withdrawal | 0 | 0

11. Secondary Outcome: Number of Patients With Elevated IFN alpha2b Protein Levels in Urine
Description: The levels of urine IFN alpha2b protein as measured by ELISA were measured in all patients on the initial day of dosing Day 1 (pre-dose) and at Day 2, Day 4, Day 12, and for patients that did not have recurrence of HGD and received a second dose at Day 91 (pre-dose), Day 92, Day 94, and Day 103.
Time Frame: 103 Days
Population: Data are reported as the number of patients with elevated levels of IFN alpha2b levels in urine.
Measure: Count of Participants; unit: Participants
Arm/Group | rAd-IFN Dose 1x10^11vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants
  Pre-Dose Day 1: number analyzed (Participants) | 21 | 18
  Pre-Dose Day 1 | 0 | 0
  Day 2: number analyzed (Participants) | 21 | 18
  Day 2 | 21 | 18
  Day 4 | 17 | 18
  Day 12: number analyzed (Participants) | 20 | 19
  Day 12 | 1 | 6
  Pre-Dose Day 91: number analyzed (Participants) | 10 | 13
  Pre-Dose Day 91 | 0 | 0
  Day 92: number analyzed (Participants) | 10 | 11
  Day 92 | 8 | 9
  Day 94: number analyzed (Participants) | 10 | 12
  Day 94 | 5 | 3
  Day 103: number analyzed (Participants) | 8 | 13
  Day 103 | 0 | 0

12. Secondary Outcome: Number of Patients With Elevated Levels of Anti-IFN alpha2b Antibodies in Serum
Description: The levels of serum anti-IFN alpha2b antibodies as measured by ELISA were determined in all patients on the initial day of dosing (Pre-Dose Day 1), at Day 12, and for patients that were free of High-Grade disease recurrence and received subsequent doses at Day 180 (pre-dose), Day 270 (pre-dose), and Day 360 or Withdrawal.
Time Frame: 360 Days
Population: Data are reported at Number of Patients with a Positive Titre.
Measure: Count of Participants; unit: Participants
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Number analyzed (Participants) | 21 | 19
Participants
  Pre-Dose Day 1 | 0 | 0
  Day 12: number analyzed (Participants) | 20 | 17
  Day 12 | 0 | 1
  Pre-Dose Day 180: number analyzed (Participants) | 8 | 9
  Pre-Dose Day 180 | 0 | 0
  Pre-Dose Day 270: number analyzed (Participants) | 8 | 9
  Pre-Dose Day 270 | 0 | 0
  Day 360 or Withdrawal: number analyzed (Participants) | 21 | 15
  Day 360 or Withdrawal | 0 | 0

13. Secondary Outcome: Number of Patients With Elevated Levels of Anti-Adenovirus Type 5 Antibodies in Serum.
Description: The levels of serum anti-adenovirus type 5 antibodies as measured by ELISA were determined in all patients on the initial day of dosing (Pre-Dose Day 1), at Day 12, and for patients that were free of High-Grade disease recurrence and received subsequent subsequent doses at Day 180 (pre-dose), Day 270 (pre-dose), and Day 360 or Withdrawal.
Time Frame: 360 Days
Population: Data are reported at Number of Patients with a Positive Titer.
Measure: Count of Participants; unit: Participants
Groups:
- rAd-IFN Dose 3x10^11vps/mL: Patients were randomly assigned to the 3x10^11 vps/ml rAd-IFN/Syn3 arm.
Arm/Group | rAd-IFN Dose 1x10^11vps/ml | rAd-IFN Dose 3x10^11vps/mL
Number analyzed (Participants) | 21 | 19
Participants
  Pre-Dose Day 1: number analyzed (Participants) | 21 | 18
  Pre-Dose Day 1 | 0 | 0
  Day 12: number analyzed (Participants) | 20 | 17
  Day 12 | 2 | 1
  Pre-Dose Day 180: number analyzed (Participants) | 8 | 9
  Pre-Dose Day 180 | 6 | 6
  Pre-Dose Day 270: number analyzed (Participants) | 8 | 9
  Pre-Dose Day 270 | 6 | 5
  Day 360 or Withdrawal: number analyzed (Participants) | 21 | 15
  Day 360 or Withdrawal | 12 | 7

ADVERSE EVENTS:
Time Frame: From dosing day 1 up to 12 months
Groups:
- rAd-IFN Dose 1x10^11 Vps/ml: Patients were randomized to the 1x10^11 vps/ml INSTILADRIN arm.
- rAd-IFN Dose 3x10^11vps/ml: Patients were randomized the 3x10^11 vps/ml INSTILADRIN arm.
Arm/Group | rAd-IFN Dose 1x10^11 Vps/ml | rAd-IFN Dose 3x10^11vps/ml
Serious Adverse Events (participants affected / at risk) | 3/21 | 2/19
Other Adverse Events (participants affected / at risk) | 20/21 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAd-IFN Dose 1x10^11 Vps/ml (N=21) | rAd-IFN Dose 3x10^11vps/ml (N=19)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Secondary to carotid artery stenosis - not related to drug; grade 3; resolved
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — not related to drug; grade 3; resolved
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — related to drug; grade 3; resolved
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) — Coronary artery blockage; not related to drug; grade 3; resolved
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) — Right carotid blockade
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Left renal pelvis tumor - not related to drug; grade 3; resolved
Nephroureterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — not related to drug; grade 3; resolved
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) — delayed return of bowel function; not related to drug; grade 3; resolved
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — worsening of back pain; related to disease; not related to drug; grade 3; resolved
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) — acute renal failure, pre-renal (dehydration); related to drug; grade 3; resolved
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAd-IFN Dose 1x10^11 Vps/ml (N=21) | rAd-IFN Dose 3x10^11vps/ml (N=19)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Oesophageal Dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 7 (7)
Facial Pain (General disorders) | 0 (0) | 1 (1)
Fatique (General disorders) | 6 (6) | 7 (7)
Feeling Cold (General disorders) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 2 (2) | 0 (0)
Infusion Site Reactions (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 6 (6)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gasteroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Nasophanryngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 5 (5)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Creatinine Increase (Investigations) | 0 (0) | 1 (1)
Glycosylated Hemoglobin Increase (Investigations) | 1 (1) | 0 (0)
pH Urine Decreased (Investigations) | 0 (0) | 1 (1)
Urine Output DeEcreased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid Retention (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oedemia Peripheral (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertrebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo Maligno Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Restless Leg Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Change (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder Discomfort (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Pain (Renal and urinary disorders) | 0 (0) | 3 (3)
Bladder Perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 9 (9) | 7 (7)
Hematuria (Renal and urinary disorders) | 5 (5) | 5 (5)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 10 (10) | 6 (6)
Nocturia (Renal and urinary disorders) | 5 (5) | 5 (5)
Pollakiuria (Renal and urinary disorders) | 6 (6) | 5 (5)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine Flow Decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatic Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythemia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nephroureterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Eye Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will complete its review within the review period and will have authority to require that the Institution and/or Investigator delete from the disclosure of any reference to Confidential Information, other than results.